CLINICAL TRIAL: NCT06389318
Title: Comparison Between Buccal Midazolam Versus Intranasal Dexmedetomidine Plus Oral Chloral Hydrate in Reducing Parental Separation Anxiety in Children Undergoing Inguinal Hernia Repair: A Randomized Clinical Trial
Brief Title: Buccal Midazolam Versus Intranasal Dexmedetomidine Plus Oral Chloral Hydrate in Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ramy Mousa, Anesthesia and surgical ICU department, Faculty of Medicine, Benha University, Egypt, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC 29-11-2023
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-04

CONDITIONS: Inguinal Hernia Repair
Keywords: Midazolam; Dexmedetomidine; Chloral Hydrate
MeSH Terms: interventions — Chloral Hydrate

STUDY DESIGN:
Intervention Model Description: Group A (40 patients): Children received oral placebo syrup, Group B (40 patients): Children received oral chloral hydrate (Chloral Hydrate mixture)
Who Masked: Participant, Care Provider
Masking Description: Both participant and the care-provider in this trial were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- buccal midazolam group (Experimental): Children received oral placebo syrup, intranasal 0.9 % normal saline at 0.03 ml/kg and buccal midazolam at 0.1 mg/ kg mixed with simple syrup
  Interventions: Drug: buccal midazolam +oral placebo syrup
- oral chloral hydrate and intranasal dexmedetomidine group (Experimental): Children received oral chloral hydrate (Chloral Hydrate mixture, concentration at 0.5gm/5ml, 250 ml bottle, at 50 mg /kg, intranasal dexmedetomidine at 2 μg/kg and buccal normal saline.
  Interventions: Drug: oral chloral hydrate,intranasal dexmedetomidine and buccal normal saline

INTERVENTIONS:
Drug: buccal midazolam +oral placebo syrup — Children received oral chloral hydrate (Chloral Hydrate mixture, concentration at 0.5gm/5ml, 250 ml bottle, prepared at abo Elreesh pharmacy, Elmoneerah , Egypt) at 50 mg /kg, intranasal dexmedetomidine at 2 μg/kg and buccal normal saline. Dexmedetomidine used was preservative-free dexmedetomidine (Precedex, 2ml ampoule,100 ug /ml, Hospira, Inc, Rocky Mount, USA) in a concentration of 100 μg/mL. Undiluted drug was withdrawn into a 1 mL tuberculin syringe.
  Other Names: Group A
  Arms: buccal midazolam group
Drug: oral chloral hydrate,intranasal dexmedetomidine and buccal normal saline — Children received oral chloral hydrate (Chloral Hydrate mixture, concentration at 0.5gm/5ml, 250 ml bottle, prepared at abo Elreesh pharmacy, Elmoneerah , Egypt) at 50 mg /kg, intranasal dexmedetomidine at 2 μg/kg and buccal normal saline. Dexmedetomidine used was preservative-free dexmedetomidine (Precedex, 2ml ampoule,100 ug /ml, Hospira, Inc, Rocky Mount, USA) in a concentration of 100 μg/mL. Undiluted drug was withdrawn into a 1 mL tuberculin syringe.
  Other Names: Group B
  Arms: oral chloral hydrate and intranasal dexmedetomidine group

SUMMARY:
Inguinal hernia surgery is one of the most common surgical procedures in early infancy. Preoperative anxiety remains a vexing issue, and it exists in nearly 50% of pediatric patients

DETAILED DESCRIPTION:
Inguinal hernia surgery is one of the most common surgical procedures in early infancy. Preoperative anxiety remains a vexing issue, and it exists in nearly 50% of pediatric patients.

The administration of sedatives to a child before entering a surgical room is the most common way of reducing the child's distress and allows the child to undergo smooth anesthesia induction.

Chloral hydrate is a widely used sedative for young children undergoing imaging studies, with a high success rate.

Dexmedetomidine is a highly selective alpha-2 agonist for paediatric sedation. It produces sedation like natural non-rapid eye movement sleep and has respiratory-sparing effect.

ELIGIBILITY:
Inclusion Criteria:

* aged 2 to 7
* American Society of Anaesthesiology (ASA) І and П scheduled for inguinal hernia repair

Exclusion Criteria:

* sensitivity to dexmedetomidine or midazolam,
* infection of the upper respiratory tract,
* severe liver or kidney disease, organ dysfunction,
* cardiac arrhythmia or congenital heart disease

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-03-26 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Ramsay sedation score | RSSs were recorded just immediately before and at 10 minutes , 20 minutes , 30 minutes after dosing
  The scoring criteria were as follows: (1) patient shows anxiety and restlessness; (2) patient is cooperative, oriented, and quiet; (3) patient is responsive to instructions; (4) patient shows somnolence and responsive to the tapping of the glabella or to loud auditory stimuli; (5) patient shows somnolence and unresponsive to the tapping of the glabella or to loud auditory stimuli; and (6) patient shows somnolence without any response.

SECONDARY OUTCOMES:
Parental separation anxiety scale | Preoperatively
  Parental separation anxiety scale was determined when the child was separated from the parents according to four levels:
  1. easy to separate
  2. sobbing but easy to cease
  3. crying loudly and difficult to stop but without holding the parents and not letting them go
  4. crying loudly and holding the parents and not willing to let them go. PSAS scores of 1 and 2 were considered "successful separation from parents

CONTACTS AND LOCATIONS:
Overall Officials: Ramy Saleh, MD, Principal Investigator — Anesthesia and surgical ICU department, Faculty of Medicine, Benha University, Egypt
Locations (1):
- Benha University, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: No
The data will be available upon reasonable request from the principle investigator